CLINICAL TRIAL: NCT05128292
Title: Role of the NLRP3 Inflammasome Activation, Mitochondrial Biogenesis, and Immunoinflammatory Response After Oral Coenzyme Q10 Plus Selenium Supplementation in Individuals With Myalgic Encephalomyelitis/Chronic Fatigue Syndrome
Brief Title: Effect of CoQ10 Plus Selenium Supplementation on Clinical Outcomes and Biochemical Markers in ME/CFS (CoSeME Study)
Acronym: CoSeME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Pharma Nord (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR(AG)233(2016)
Record Dates: First submitted 2021-11-05; First posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Myalgic Encephalomyelitis
Keywords: fatigue; Coenzyme Q10; selenium; sleep disturbances; biomarkers; myalgic encephalomyelitis; chronic fatigue syndrome
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Fatigue; Parasomnias | interventions — coenzyme Q10; Selenium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CoQ10 plus selenium (Experimental): Nutraceutical intervention:
  400 mg/day CoQ10 soft gel capsula (Bio-Quinone active 100 mg b.i.d) plus 200 microgram organic selenium yeast tablet (SelenoPrecise 100 microgram b.i.d.) over 8 weeks
  Interventions: Dietary Supplement: CoQ10 plus Selenium

INTERVENTIONS:
Dietary Supplement: CoQ10 plus Selenium — 400 mg/day CoQ10 soft gel capsula (Bio-Quinone active 100 mg b.i.d) plus 200 microgram organic selenium yeast tablet (SelenoPrecise 100 microgram b.i.d.) over 8 weeks

SUMMARY:
In recent years, it has been suggested that nutritional deficiencies may be of causal relevance in individuals with ME/CFS. These include deficiencies of vitamins and trace elements. It is likely that the observed nutritional deficiencies contribute to the core symptoms of the disease. Coenzyme Q10 (CoQ10) has been studied as an alternative and complementary therapy in ME/CFS for fatigue, pain, tiredness, neurocognitive impairment, and sleep problems. This demonstrates how alterations in energy metabolism, mitochondrial dysfunction, oxidative stress, imbalance of the immune-inflammatory response, and activation of the NLRP3 inflammasome are likely consequences of low levels of CoQ10 and selenium, which are related to the main symptoms in ME/CFS. Hypothesis: CoQ10 and selenium levels are decreased in ME/CFS patients. A natural therapeutic alternative in the treatment of common symptoms in ME/CFS could be the oral CoQ10 (Ubiquinone) plus selenium supplementation to module redox status and inflammation response in ME/CFS. Aims: To evaluate the efficacy of oral Ubiquinone + selenium supplementation on clinical outcome and circulating biomarkers in ME/CFS. We enrolled 42 ME/CFS patients diagnosed according to the 1994 CDC/Fukuda criteria who have received oral treatment of 400 mg Ubiquinone + 200 microgram selenium daily for 8 weeks. Demographic, clinical characteristics and laboratory variables, and validated outcome measures to perceived fatigue, sleep disturbances, and quality of life will be also evaluated. In addition, plasma biomarkers related to oxidative stress status (total antioxidant capacity and lipoperoxide levels), inflammatory response (pro-and anti-inflammatory cytokines), and cardiovascular dysfunction (FGF-21 and NT-proBNP) will be assayed.

ELIGIBILITY:
Inclusion Criteria:

* Patients were potentially eligible if they were female, aged 18 years or older, and had a confirmed diagnosis of ME/CFS by a specialist according to the 1994 CDC/Fukuda criteria

Exclusion Criteria:

* Exclusion criteria were those with any significant active fatiguing medical disorder (thyroid-related disorders, sleep apnea, narcolepsy, medication side-effects, heart diseases, iron deficiency anemia), previous diagnosis not unequivocally resolved (chronic hepatitis, malignancy), autoimmune disorders, history of past/current neuropsychiatric disorders (major depressive disorder, psychotic or melancholic features, bipolar disorder, schizophrenia, delusional disorder, dementias, anorexia nervosa, and bulimia nervosa), and participation in another clinical trial of the same or different nature within 30 days prior to study inclusion; inability (in the opinion of the investigator) to follow the instructions or to complete the treatment satisfactorily; failure to provide signed informed consent; use of certain drugs and supplements that might influence outcome measures in the last 90 days or whose withdrawal might be a relevant problem, anticoagulant treatment, pregnancy or breast-feeding, smoking habits, alcohol intake or substance abuse, strong hormone-related medications, and obesity.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Fatigue perception assessed through FIS-40 questionnaire | 8 weeks
  FIS-40 self-reported questionnaire: Change of fatigue perception from baseline will be assessed.

SECONDARY OUTCOMES:
Sleep disturbances evaluated through PSQI | 8 weeks
  Change of sleep problems from baseline will be assessed.
Health-related quality of life assessed by SF-36 | 8 weeks
  Change of quality of life (SF-36) from baseline will be assessed.
Measurement of biomarkers of redox status. | 8 weeks
  Change of the circulating biomarker levels of oxidative stress (malondialdehydes and total antioxidant capacity) from baseline will be measured.
Measurement of biomarkers of inflammatory immune response. | 8 weeks
  Change of the circulating biomarker levels of inflammatory cytokines (IL-1 beta, IL-6, IL-8, IL-10, TNF-alpha, and C-reactive protein) from baseline will be measured.
Measurement of biomarkers of cardiovascular risk. | 8 weeks
  Change of the circulating biomarker levels of cardiovascular function (FGF-21 and NT-proBNP) from baseline will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: José Alegre, MD, PhD, Principal Investigator — Vall d'Hebron University Hospital
Locations (1):
- Vall d'Hebron University Hospital, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bjorklund G, Dadar M, Pen JJ, Chirumbolo S, Aaseth J. Chronic fatigue syndrome (CFS): Suggestions for a nutritional treatment in the therapeutic approach. Biomed Pharmacother. 2019 Jan;109:1000-1007. doi: 10.1016/j.biopha.2018.10.076. Epub 2018 Nov 5. PMID 30551349
- [Background] Morris G, Puri BK, Walker AJ, Maes M, Carvalho AF, Walder K, Mazza C, Berk M. Myalgic encephalomyelitis/chronic fatigue syndrome: From pathophysiological insights to novel therapeutic opportunities. Pharmacol Res. 2019 Oct;148:104450. doi: 10.1016/j.phrs.2019.104450. Epub 2019 Sep 8. PMID 31509764
- [Background] Testai L, Martelli A, Flori L, Cicero AFG, Colletti A. Coenzyme Q10: Clinical Applications beyond Cardiovascular Diseases. Nutrients. 2021 May 17;13(5):1697. doi: 10.3390/nu13051697. PMID 34067632
- [Background] Fukuda S, Nojima J, Kajimoto O, Yamaguti K, Nakatomi Y, Kuratsune H, Watanabe Y. Ubiquinol-10 supplementation improves autonomic nervous function and cognitive function in chronic fatigue syndrome. Biofactors. 2016 Jul 8;42(4):431-40. doi: 10.1002/biof.1293. Epub 2016 Apr 29. PMID 27125909
- [Background] Maes M, Mihaylova I, Kubera M, Uytterhoeven M, Vrydags N, Bosmans E. Coenzyme Q10 deficiency in myalgic encephalomyelitis/chronic fatigue syndrome (ME/CFS) is related to fatigue, autonomic and neurocognitive symptoms and is another risk factor explaining the early mortality in ME/CFS due to cardiovascular disorder. Neuro Endocrinol Lett. 2009;30(4):470-6. PMID 20010505
- [Background] Nacul L, Authier FJ, Scheibenbogen C, Lorusso L, Helland IB, Martin JA, Sirbu CA, Mengshoel AM, Polo O, Behrends U, Nielsen H, Grabowski P, Sekulic S, Sepulveda N, Estevez-Lopez F, Zalewski P, Pheby DFH, Castro-Marrero J, Sakkas GK, Capelli E, Brundsdlund I, Cullinan J, Krumina A, Bergquist J, Murovska M, Vermuelen RCW, Lacerda EM. European Network on Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (EUROMENE): Expert Consensus on the Diagnosis, Service Provision, and Care of People with ME/CFS in Europe. Medicina (Kaunas). 2021 May 19;57(5):510. doi: 10.3390/medicina57050510. PMID 34069603
- [Result] Castro-Marrero J, Cordero MD, Segundo MJ, Saez-Francas N, Calvo N, Roman-Malo L, Aliste L, Fernandez de Sevilla T, Alegre J. Does oral coenzyme Q10 plus NADH supplementation improve fatigue and biochemical parameters in chronic fatigue syndrome? Antioxid Redox Signal. 2015 Mar 10;22(8):679-85. doi: 10.1089/ars.2014.6181. Epub 2014 Dec 18. PMID 25386668
- [Result] Campagnolo N, Johnston S, Collatz A, Staines D, Marshall-Gradisnik S. Dietary and nutrition interventions for the therapeutic treatment of chronic fatigue syndrome/myalgic encephalomyelitis: a systematic review. J Hum Nutr Diet. 2017 Jun;30(3):247-259. doi: 10.1111/jhn.12435. Epub 2017 Jan 22. PMID 28111818
- [Result] Castro-Marrero J, Saez-Francas N, Segundo MJ, Calvo N, Faro M, Aliste L, Fernandez de Sevilla T, Alegre J. Effect of coenzyme Q10 plus nicotinamide adenine dinucleotide supplementation on maximum heart rate after exercise testing in chronic fatigue syndrome - A randomized, controlled, double-blind trial. Clin Nutr. 2016 Aug;35(4):826-34. doi: 10.1016/j.clnu.2015.07.010. Epub 2015 Jul 17. PMID 26212172
- [Result] Castro-Marrero J, Segundo MJ, Lacasa M, Martinez-Martinez A, Sentanes RS, Alegre-Martin J. Effect of Dietary Coenzyme Q10 Plus NADH Supplementation on Fatigue Perception and Health-Related Quality of Life in Individuals with Myalgic Encephalomyelitis/Chronic Fatigue Syndrome: A Prospective, Randomized, Double-Blind, Placebo-Controlled Trial. Nutrients. 2021 Jul 30;13(8):2658. doi: 10.3390/nu13082658. PMID 34444817
- [Result] Castro-Marrero J, Cordero MD, Saez-Francas N, Jimenez-Gutierrez C, Aguilar-Montilla FJ, Aliste L, Alegre-Martin J. Could mitochondrial dysfunction be a differentiating marker between chronic fatigue syndrome and fibromyalgia? Antioxid Redox Signal. 2013 Nov 20;19(15):1855-60. doi: 10.1089/ars.2013.5346. Epub 2013 May 29. PMID 23600892
- [Result] Maksoud R, Balinas C, Holden S, Cabanas H, Staines D, Marshall-Gradisnik S. A systematic review of nutraceutical interventions for mitochondrial dysfunctions in myalgic encephalomyelitis/chronic fatigue syndrome. J Transl Med. 2021 Feb 17;19(1):81. doi: 10.1186/s12967-021-02742-4. PMID 33596913